CLINICAL TRIAL: NCT05681650
Title: Phase I/II Clinical Trial of HER2 Targeted HypoSti.CAR-T Cells in Treating Patients With HER2 Positive Local Advanced or Metastatic Solid Tumors
Brief Title: HER2 Targeted HypoSti.CAR-T Cells in HER2 Positive Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Fudan University (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-076
Record Dates: First submitted 2022-12-27; First posted 2023-01-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: HER2 Positive Advanced Solid Tumors
MeSH Terms: interventions — Albumin-Bound Paclitaxel; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HypoSti.CAR-HER2 T cells (Experimental): Enrolled participants will be given a preconditioning regimen consisted of albumin-bound paclitaxel, cyclophosphamide and/or fludarabine before the infusion of HypoSti.CAR-HER2 T cells. Fludarabine will be administered only before the first dose infusion, and will not be administered before the secondary or multiple doses of HypoSti.CAR-HER2 T cell infusion.
  Interventions: Biological: HypoSti.CAR-HER2 T cells; Drug: Albumin-bound paclitaxel; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: HypoSti.CAR-HER2 T cells — Dose escalation: dose -1 (1×10^6 cells/kg) ,dose 1 (3×10^6 cells/kg) , dose 2 (6×10^6 cells/kg), dose 3 (1×10^7 cells/kg), dose 4 (1.5×10^7 cells/kg). Dose expansion: RP2D
Drug: Albumin-bound paclitaxel — Administered intravenously at dose of 100-200mg/m2 on day -5
Drug: Cyclophosphamide — Administered intravenously at a total dose of 15-30mg/kg on day -3 and day-2
Drug: Fludarabine — Administered intravenously at dose of 30mg/m2/d on day -3 and day -2 only in the first infusion of HypoSti.CAR-HER2 T cells

SUMMARY:
Chimeric antigen receptor modified T (CAR-T) cell therapy still has multiple difficulties in solid tumors, such as absence of tumor specific antigens, complex immunosuppressive tumor microenvironment, and tumor heterogeneity. In this study, investigators developed a novel hypoxia-stimulated CAR expression system (HypoSti.CAR) that could enable CAR-T cell effectively expand and survive in hypoxic tumor microenvironment. After accomplishment of animal model verification, investigators conduct this clinical trial in order to assess the in vivo safety, feasibility and efficacy of HypoSti.CAR-HER2 T cells in HER2 antigen positive advanced solid tumors.

DETAILED DESCRIPTION:
Currently, chimeric antigen receptor modified T (CAR-T) cell therapy has achieved a series of achievements in hematological malignancies, however, it still has to face plenty of obstacles in more bulky solid tumors, such as absence of tumor specific antigens, complex immunosuppressive tumor microenvironment, and tumor heterogeneity, which may taken together to restrict the efficacy of CAR-T cells in eliminating solid tumors. Previous studies found that intratumoral hypoxic microenvironment facilitated the development and metastasis of tumor cells. Meanwhile, it was difficult for cytotoxic T cells including CAR-T cells to survive and expand in such a hypoxic microenvironment.

In this study, investigators developed a novel hypoxia-stimulated CAR expression system (HypoSti.CAR) that could enable CAR-T cell effectively expand and survive in hypoxic tumor microenvironment,which has been demonstrated in animal models. Based on the preclinical data, investigators will further conduct this clinical trial in order to test the potential of this novel system targeting HER2 antigen in vivo. In dose escalation period, at least 9 eligible patients will be enrolled and receive 5 doses of HypoSti.CAR-HER2 T cell therapy (1 × 10^6 cells/kg, 3 × 10^6 cells/kg, 6 × 10^6 cells/kg,1 × 10^7 cells/kg, 1.5 × 10^7 cells/kg) according to the "3+3" principle. In dose expansion period, additional 10 to 21 patients will be enrolled to receive HypoSti.CAR-HER2 T cell therapy at dose of recommended phase 2 dose (RP2D), which is determined by data from dose escalation period, including occurrence of dose limiting toxicities (DLT), pharmacokinetics/pharmacodynamics, efficacy and other parameters, to furtherly evaluate the safety and efficacy profiles of HypoSti.CAR-HER2 T cell therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age from 18 to 75 years with estimated life expectancy >3 months.
* 2. Histopathological confirmed advanced or metastatic solid tumors failed to at least first-line treatment or initially diagnosed advanced/metastatic solid tumors that have no NCCN guideline recommended standard first-line therapy. HER2 antigen expression percentage ≥ 30%.
* 3. Have at least one measurable target lesion.
* 4. Fresh solid tumor samples or formalin-fixed paraffin embedded tumor archival samples within 6 months are necessary; Fresh tumor samples are preferred. Subjects are willing to accept tumor rebiopsy in the process of this study.
* 5. Previous treatment must be completed for more than 4 weeks prior to the enrollment of this study, and subjects have recovered to <= grade 1 toxicity.
* 6. Have an Eastern Cooperative Oncology Group performance status (ECOG) of 0 or 2 at the time of enrollment.
* 7. Have adequate organ function, which should be confirmed within 2 weeks prior to the first dose of study drugs.
* 8. Previous treatment with anti-PD-1/PD-L1 antibodies are allowed.
* 9. Ability to understand and sign a written informed consent document.
* 10. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, and up to 90 days after the last dose of the drug.

Exclusion Criteria:

* 1. Active, known or suspected autoimmune diseases.
* 2. Known brain metastases or active central nervous system (CNS). Subjects with CNS metastases who were treated with radiotherapy for at least 3 months prior to enrollment, have no central nervous symptoms and are off corticosteroids, are eligible for enrollment, but require a brain MRI screening.
* 3. Subjects are being treated with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrollment.
* 4. History of severe hypersensitive reactions to other monoclonal antibodies.
* 5. History of allergy or intolerance to study drug components.
* 6. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
* 7. History or concurrent condition of interstitial lung disease of any grade or severely impaired pulmonary function.
* 8. Uncontrolled intercurrent illness, including ongoing or active systemic infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (excluding insignificant sinus bradycardia and sinus tachycardia) or psychiatric illness/social situations and any other illness that would limit compliance with study requirements and jeopardize the safety of the patient.
* 9. History of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS).
* 10. Pregnant or breast-feeding. Women of childbearing potential must have a pregnancy test performed within 7 days before the enrollment, and a negative result must be documented.
* 11. Previous or concurrent cancer within 3 years prior to treatment start EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer, superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
* 12. Vaccination within 30 days of study enrollment.
* 13. Active bleeding or known hemorrhagic tendency.
* 14. Subjects with unhealed surgical wounds for more than 30 days.
* 15. Being participating any other trials or withdraw within 4 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment related adverse events | Up to 12 months following the infusion of HypoSti.CAR-HER2 T cells
  Treatment related adverse events are defined as any medical events since the initiation of preconditioning chemotherapy. Adverse events will be graded by CTCAE V5.0
Incidence of dose limiting toxicities (DLTs) | Up to 28 days following the infusion of HypoSti.CAR-HER2 T cells
  Dose limiting toxicities are defined as HypoSti.CAR-HER2 T cell related adverse events within the first 28 days that meet the following criteria: grade 3 or higher CRS or CRES, grade 3 or higher cutaneous/ mucosal toxicity, and any other grade 4 toxicities.
Determination of the maximum tolerated dose (MTD) | Up to 28 days following the infusion of HypoSti.CAR-HER2 T cells
  Maximum tolerated dose is defined as the highest dose that is less than or equal to 2 DLT among 6 subjects.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 3 years
  Objective response rate is defined as complete response (CR) or partial response (PR) by RECIST 1.1or iRECIST
Time to response (TTR) | Up to 3 years
  Time to response is defined as the time from HypoSti.CAR-HER2 T cell infusion to first assessed CR or PR by investigators according to RECIST 1.1or iRECIST.
Duration of response (DOR) | Up to 3 years
  Duration of response is defined as the time from objective response (OR) until documented tumor progression date among responders.
Progression Free Survival (PFS) | Up to 3 years
  Progression Free Survival is defined as the time from HypoSti.CAR-HER2 T cell infusion to documented disease progression or death.
Overall Survival (OS) | Up to 3 years
  Overall Survival is defined as the time from HypoSti.CAR-HER2 T cell infusion to the date of death.
Number and copy number of HypoSti.CAR-HER2 T cell | Up to 3 years
  Number and copy number of HypoSti.CAR-HER2 T cell are assessed by number in peripheral blood and tumor tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Jianqing Xu, PhD, Study Director — Fudan University
Locations (1):
- Kaichao Feng, Beijing, Beijing Municipality, China